CLINICAL TRIAL: NCT01971866
Title: Improving Safety and Accuracy of Proton Therapy by Use of Camera-Based Patient Localization System
Brief Title: Camera Based System to Monitor Patient Movement During Radiation Treatment
Acronym: DS02
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment, feasibility issues
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFPTI 1215-DS02
Record Dates: First submitted 2013-10-17; First posted 2013-10-29 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Set up and Monitoring of Patients Receiving Proton Radiation
Keywords: Proton radiation; AlignRT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to investigate the advantages of using AlignRT, a commercially available, FDA approved camera-based imaging system for proton therapy patients prior to and during their radiation treatment delivery.

ELIGIBILITY:
Inclusion Criteria:

Patients with tumors of the brain, head and neck, thorax, upper abdomen, posterior spine/sacrum and extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing proton radiation therapy at UFPTI
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Paired difference between image accuracy plan data from the AlignRT system compared to the current x-ray based imaging system. | 3 months
  Enrollment and analysis will be restricted to adult patients with tumors of the brain, head and neck region, thorax, upper abdomen, or posterior spine/sacrum. Primary outcome will be analyzed by paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Mamalui-Hunter, PhD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States